CLINICAL TRIAL: NCT00527189
Title: Which Measures of Balance Best Discriminate Balance Impairment and Falls Risk in People With Lower Limb Arthritis, and Can These be Improved With Exercise?
Brief Title: Balance Impairment and Falls Risk in People With Lower Limb Arthritis, and Can These be Improved With Exercise?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Ageing Research Institute, Australia (Other)
Collaborators: Melbourne Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98765
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Arthritis
Keywords: Arthritis; Exercise; Balance - Postural Control
MeSH Terms: conditions — Arthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Balance Exercises — Home based balance exercises based on Otago Exercise programme

SUMMARY:
Arthritis has been reported as a risk factor for falls. Few studies have investigated the effect of balance training on balance performance in women with lower limb arthritis. The aim of this study was to evaluate the effectiveness of a four-month individualised home exercise programme in improving gait stability and balance for women with arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb osteoarthritis or lower limb rheumatoid arthritis

Exclusion Criteria:

Participants were excluded if they:

* Did not have lower limb arthritis,
* Were bed bound,
* Had additional co-morbidities that confer risk of falls (such as Parkinson's disease, stroke, multiple sclerosis, history of cardiac syncope, epilepsy),
* Had undergone lower limb surgery within the previous twelve months, and/or
* Had synvisc or a corticosteroid injection within the last six months.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Falls Risk Human Activity Profile Confidence Balance Measures Gait Measures

CONTACTS AND LOCATIONS:
Overall Officials: Keith Hill, PhD, Principal Investigator — National Ageing Research Institue, Australia
Locations (1):
- National Ageing Research Institute, Melbourne, Victoria, Australia